CLINICAL TRIAL: NCT03883646
Title: Mindfulness for Alcohol Abusing Offenders
Acronym: MIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Mind Research Network (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Kent Kiehl, Professor of Psychology, Neuroscience and Law, Executive Science Officer, The Mind Research Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18114
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Abuse; Criminal Behavior
MeSH Terms: conditions — Alcoholism; Criminal Behavior | interventions — Mindfulness; Secondary Prevention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness (Experimental): Mindfulness
  Interventions: Behavioral: Mindfulness
- Relapse Prevention (Experimental)
  Interventions: Behavioral: Relapse Prevention
- Waitlist Control (No Intervention)
- Treatment as Usual (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness-based Relapse Prevention. Guided meditation/discussion (Group sessions).
  Arms: Mindfulness
Behavioral: Relapse Prevention — Relapse Prevention. Cognitive behavioral principles/strategies (Group sessions).
  Arms: Relapse Prevention

SUMMARY:
Over half of state and federal prisoners meet clinical criteria for alcohol abuse or dependence, and after release from prison, over three-quarters of offenders are re-arrested within five years. Thus, there is a critical need for more effective interventions that could help disrupt this insidious cycle of alcohol abuse, criminal behavior, and incarceration. This project will support the development and evaluation of a mindfulness intervention for female prison inmates that will target key neuropsychological vulnerabilities that are associated with relapse and recidivism.

DETAILED DESCRIPTION:
The pernicious link between substance abuse and criminal behavior imposes major costs to society, totaling billions of dollars in the U.S. annually. There is a critical need for more effective interventions to counteract the high rates of relapse and recidivism in alcohol and substance abusing criminal offenders. Periods of offender incarceration provide a unique opportunity to develop and deploy such interventions. Progress in intervention development could be achieved by targeting specific cognitive and affective vulnerabilities that are common among substance abusing criminal offenders. Preliminary studies suggest that meditative or mindfulness interventions may confer significant psychological and behavioral benefits to inmates. However, the mechanisms and extent of intervention efficacy are unclear, as these previous studies have been beset by a number of methodological limitations. Moreover, to date no study has examined the neurobiological mechanisms that relate to treatment success in this population. NIAAA has recently made a program call to address these issues (PA-15-299). Here we answer this program call and propose to undertake a rigorous and comprehensive longitudinal study of mindfulness treatment of alcohol and substance use disorders among female inmates. This project will randomly assign over 400 female inmates to a mindfulness or relapse prevention training course, and both will be compared against a no treatment control. The mindfulness intervention will be tailored to address two key neuropsychological deficits in alcohol abusing criminal offenders: impulsivity and craving. We will test hypotheses about the neural changes over time with treatment to elucidate mechanisms of change. We will obtain estimates of "real-world" efficacy of the intervention by collecting outcome measures in prison (conduct reports) and following release (alcohol use relapse and antisocial behavior). This project takes advantage of a unique, longstanding partnership between the research team and the states of New Mexico and Wisconsin Correction Departments that allows collection of comprehensive assessment data from inmates during incarceration, including brain imaging data with a mobile MRI scanner, as well as access to post-release outcomes and relapse data. Completion of these aims is a critical step for implementing and evaluating a promising mindfulness intervention for this high-risk population. The proposed research will also begin to elucidate the psychological and neurobiological mechanisms of the treatment. These results will thus significantly advance a program of research seeking to translate the growing knowledge of neuropsychological deficits into more targeted and effective treatments for alcohol and substance abuse problems in criminal offenders.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Alcohol Use Disorder
* Female (biological sex at birth)
* Time to release from incarceration > 3 months
* 5th grade or higher reading level
* Able to speak and understand English

Exclusion Criteria:

* Uncorrectable auditory or visual deficits
* Intelligence Quotient score below 70
* History of dementia or other cognitive disability
* Current psychotic disorder (chronic schizophrenia or schizoaffective disorder and/or active psychotic symptoms)
* Major medical illness or Central Nervous System disease
* MRI incompatibility (e.g., metal in body)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 392 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline alcohol craving | 4 weeks, 8 weeks, and after release from incarceration (every 3 months)
  Penn Alcohol Craving Scale. 5-item, self-report measure assessing frequency, intensity, and duration of craving, and overall rating of craving for the previous week. Total score range 0-30. Higher scores indicate higher craving.
Change from baseline daily alcohol consumption | Every 3 months after release from incarceration
  Timeline Follow Back
Change from baseline temptation to drink alcohol | 4 weeks, 8 weeks, and after release from incarceration (every 3 months)
  Abstinence Self-Efficacy Scale. 40-item, self-report measure assessing how tempted the participant found themselves to drink under various circumstances. Total score range 0-160. Higher scores indicate higher temptation to drink.
Criminal Behavior | An average of six months after release from incarceration
  Crime Inventory

CONTACTS AND LOCATIONS:
Locations (1):
- The Mind Research Network, Albuquerque, New Mexico, United States

DOCUMENTS (1):
  • Informed Consent Form (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT03883646/ICF_002.pdf